CLINICAL TRIAL: NCT00325195
Title: Randomized, Multicenter, Double-blind, Placebo-controlled Efficacy and Safety Study of 8 mg PEG-uricase in Two Dose Regimens in Hyperuricemic Subjects With Symptomatic Gout
Brief Title: Safety and Efficacy Study of PEG-uricase in the Treatment of Hyperuricemic Patients With Symptomatic Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Responsible Party: Savient Pharmaceuticals, Inc, Savient Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0405 & C0406
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Pegloticase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- q2 wks (Experimental): 8 mg pegloticase every 2 weeks
  Interventions: Biological: pegloticase
- q4 wks (Experimental): 8 mg pegloticase every 4 weeks (alternating with placebo every 4 weeks)
  Interventions: Biological: pegloticase
- placebo (Placebo Comparator): placebo every 2 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — placebo by intravenous infusion every 2 weeks
  Arms: placebo
Biological: pegloticase — 8 mg pegloticase by intravenous infusion
  Other Names: PEG-uricase; Puricase
  Arms: q2 wks; q4 wks

SUMMARY:
These are two replicate studies to evaluate the safety and efficacy of PEG (polyethylene glycol)-uricase in controlling the uric acid level in symptomatic gout patients with high uric acid levels who are unable to take standard gout therapies, or for whom those therapies have been unsuccessful in controlling their uric acid level.

DETAILED DESCRIPTION:
The primary objective of each of the studies is to demonstrate superiority in the response rate (control of uric acid levels to below 6 mg/dL) in the PEG-uricase treatment groups compared to the placebo-control group.

While reduction or resolution of tophi have been reported in the setting of prolonged urate-lowering therapy, there is photographic and additional anecdotal evidence from the Phase 2 PEG-uricase study of resolution or significant reduction of tophi after 3 months of therapy. Therefore, an assessment of changes in tophi over time will be conducted through the use of digital photographs obtained in a standardized manner from all subjects during the study. The effect on other clinical outcomes, including quality of life, health-related disability measures, gout flares and the number of swollen and tender joints will also be compared between the treatment groups and control group. Subjects will be randomized to one of the three treatment arms in a 2:2:1 ratio: 8 mg PEG-uricase every 2 weeks; 8 mg PEG-uricase every 4 weeks; or placebo. All subjects will receive an intravenous infusion (PEG-uricase or placebo) every two weeks in order to maintain the blind throughout the study. Study duration is approximately 26 weeks, including two weeks for screening and 24 weeks (6 months) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients of either gender, age 18 or older ( no upper age limit).
2. Patient is hyperuricemic: screening serum uric acid must be ≥8 mg/dL.
3. Patient has symptomatic gout (presence of at least 3 gout flares in the 18 months prior to entry, or at least one gout tophus, or gouty arthritis).
4. Conventional therapy is contraindicated or has been ineffective in this patient, i.e., patient has a history (either by medical record or patient interview) of hypersensitivity or of failure to normalize SUA with at least 3 months treatment with allopurinol at the maximum labeled dose (800 mg/dL in the U.S.), or at a medically appropriate lower dose based on dose-limiting toxicity or dose-limiting co-morbidity.
5. Patient is willing and able to give informed consent and adhere to visit/protocol schedules (informed consent must be given before the first study procedure is performed, including washout).
6. If the patient is a woman of childbearing potential, she must have had a negative screening serum pregnancy test and must use a medically approved form of birth control during her participation in the protocol. Such methods include oral, injectable or implantable contraceptives; IUDs and barrier contraceptives in combination with spermicide. (If male or surgically sterile, check N/A.)

Exclusion Criteria:

1. The patient has unstable angina.
2. The patient has uncontrolled arrhythmia.
3. The patient has non-compensated congestive heart failure.
4. The patient has uncontrolled hypertension (above 150/95).
5. The patient has a history of end stage renal disease requiring dialysis.
6. The patient has hemoglobin < 8 g/dL (males) or < 7 g/dL (females).
7. The patient is an organ transplant recipient
8. The patient has had prior treatment with PEG-uricase, or other recombinant uricase, or any concomitant therapy with a PEG-conjugated drug.
9. The patient has had a gout flare at screening that is resolved for less than one week prior to first treatment with study drug (exclusive of chronic synovitis/ arthritis).
10. The patient has glucose-6-phosphate dehydrogenase (G6PD) deficiency.
11. The patient has a history of anaphylactic reaction to a recombinant protein or porcine product, or hypersensitivity to PEG.
12. The patient is pregnant or breast feeding.
13. The patient has taken an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study.
14. The patient has a known allergy to urate oxidase or PEGylated products.
15. The patient has any other medical or psychological condition which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Savient Pharmaceuticals, Inc.
Locations (56):
- United States (50):
  - UAB Arthritis Clinical Intervention Program, Birmingham, Alabama
  - University of Arizona Arthritis Center, Tucson, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - UCSD Rheumatology Division, La Jolla, California
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - E. Robert Harris Medical Corporation, Whittier, California
  - Agilence Arthritis & Osteoporosis Medical Center, Whittier, California
  - Arthritis Associates & Osteoporosis Center of Colorado Springs, Colorado Springs, Colorado
  - Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Arthritis & Osteoporosis Treatment Center, PA, Orange Park, Florida
  - St. Petersburg Arthritis Center, St. Petersburg, Florida
  - Idaho Arthritis & Osteoporosis Center, Boise, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - The University of Chicago, Chicago, Illinois
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Peter A. Holt, M.D., Baltimore, Maryland
  - Malamet & Klein, MD, PA, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Fallon Clinic, Inc, Worcester, Massachusetts
  - Michigan Arthritis Research Center, Brighton, Michigan
  - Justus J. Fiechtner, MD, PC, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Rheumatology Associates of North Jersey, Teaneck, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - Physicians East, P.A., Greenville, North Carolina
  - Carolina Atthritis Associates, Wilmington, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - David R. Mandel, MD, Inc., Mayfield Village, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Portland Medical Associates, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Mid Atlantic Research Assoc., Philadelphia, Pennsylvania
  - Rheumatology Associates, Charleston, South Carolina
  - Piedmont Arthritis, PA, Greenville, South Carolina
  - AAMR Research Clinic, Amarillo, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
  - Arthritis & Osteoporosis Clinic Research Center of Central Texas, Waco, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
- Canada (2):
  - Manitoba Clinic, Winnipeg, Manitoba
  - St. Joseph's Health Care, London, Ontario
- Mexico (4):
  - Clinica para el Diagnostico y Tratamiento de las Enfermedades Rheumaticas, México, D.f.
  - Hospital General de mexico, México, D.f.
  - Antiguo Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco

REFERENCES:
- [Derived] Pillinger MH, Fields TR, Yeo AE, Lipsky PE. Dissociation Between Clinical Benefit and Persistent Urate Lowering in Patients with Chronic Refractory Gout Treated with Pegloticase. J Rheumatol. 2020 Apr;47(4):605-612. doi: 10.3899/jrheum.190161. Epub 2019 Jun 15. PMID 31203212
- [Derived] Johnson RJ, Choi HK, Yeo AE, Lipsky PE. Pegloticase Treatment Significantly Decreases Blood Pressure in Patients With Chronic Gout. Hypertension. 2019 Jul;74(1):95-101. doi: 10.1161/HYPERTENSIONAHA.119.12727. Epub 2019 May 13. PMID 31079535
- [Derived] Lipsky PE, Calabrese LH, Kavanaugh A, Sundy JS, Wright D, Wolfson M, Becker MA. Pegloticase immunogenicity: the relationship between efficacy and antibody development in patients treated for refractory chronic gout. Arthritis Res Ther. 2014 Mar 4;16(2):R60. doi: 10.1186/ar4497. PMID 24588936
- [Derived] Yood RA, Ottery FD, Irish W, Wolfson M. Effect of pegloticase on renal function in patients with chronic kidney disease: a post hoc subgroup analysis of 2 randomized, placebo-controlled, phase 3 clinical trials. BMC Res Notes. 2014 Jan 21;7:54. doi: 10.1186/1756-0500-7-54. PMID 24447425
- [Derived] Baraf HS, Becker MA, Gutierrez-Urena SR, Treadwell EL, Vazquez-Mellado J, Rehrig CD, Ottery FD, Sundy JS, Yood RA. Tophus burden reduction with pegloticase: results from phase 3 randomized trials and open-label extension in patients with chronic gout refractory to conventional therapy. Arthritis Res Ther. 2013 Sep 26;15(5):R137. doi: 10.1186/ar4318. PMID 24286509
- [Derived] Sundy JS, Baraf HS, Yood RA, Edwards NL, Gutierrez-Urena SR, Treadwell EL, Vazquez-Mellado J, White WB, Lipsky PE, Horowitz Z, Huang W, Maroli AN, Waltrip RW 2nd, Hamburger SA, Becker MA. Efficacy and tolerability of pegloticase for the treatment of chronic gout in patients refractory to conventional treatment: two randomized controlled trials. JAMA. 2011 Aug 17;306(7):711-20. doi: 10.1001/jama.2011.1169. PMID 21846852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rheumatology practices across the US, Canada and Mexico
Pre-assignment Details: 13 subjects were randomized but withdrew before intervention. These subjects were not part of the modified Intent to Treat Population, which included only subjects who received at least one dose of study drug.
Groups:
- q4 Wks: 8 mg pegloticase every 4 weeks (alternating with placebo infusion every 4 weeks)
- Placebo: placebo infusion every 2 weeks
Period: Randomized
Arm/Group | q2 Wks | q4 Wks | Placebo
Started | 90 | 89 | 46
Completed | 85 | 84 | 43
Not Completed | 5 | 5 | 3
Not completed — Not dosed | 5 | 5 | 3
Period: Received Intervention: ITT Population
Arm/Group | q2 Wks | q4 Wks | Placebo
Started | 85 | 84 | 43
Completed | 59 | 59 | 39
Not Completed | 26 | 25 | 4
Not completed — Adverse Event | 15 | 17 | 1
Not completed — Death | 3 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Protocol violation/non-compliance | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | q2 Wks | q4 Wks | Placebo | Total
Number analyzed (Participants) | 85 | 84 | 43 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 65 | 31 | 152
  >=65 years | 29 | 19 | 12 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (15.53) | 54.5 (13.34) | 55.4 (12.21) | 55.4 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 7 | 39
  Male | 68 | 69 | 36 | 173
Region of Enrollment [Number; unit: participants]
  United States | 73 | 77 | 39 | 189
  Canada | 1 | 1 | 1 | 3
  Mexico | 11 | 6 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Plasma Uric Acid (PUA) Responder
Description: PUA Responder was defined as a participant who achieved and maintained plasma uric acid concentrations < 6 mg/dL for at least 80% of the time during months 3 and 6 combined. Participants who withdrew from the study before month 6 were considered non-responders.
Time Frame: Months 3 and 6
Population: Modified ITT (all patients receiving at least one dose of study drug). Participants dropping out before Week 25 were imputed as Non-Responders
Measure: Number; unit: Participants
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 85 | 84 | 43
Participants | 36 | 29 | 0
Statistical Analysis 1: Comparison: q2 Wks vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: q4 Wks vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Reduction in Tophus Burden
Description: percentage of tophaceous subjects who demonstrated a complete resolution (100 % decrease in measured area or complete disappearance)of at least one tophus in the absence of other tophus progression or new tophi, as assessed by a blinded Central Reader using standardized digital photographs and image analysis software.
Time Frame: Baseline and Final Visit (6 months or LOCF)
Population: Number of participants analyzed was based upon the number of patients who had one or more tophus at Baseline, as determined by the PI, AND who had at least one follow-up assessment, with the final visit for each subject included (last observation carried forward).
Measure: Number; unit: Percent subjects with resolved tophus
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 52 | 52 | 27
Percent subjects with resolved tophus | 40 | 21 | 7
Statistical Analysis 1: Comparison: q2 Wks vs Placebo; Test type: Superiority or Other; p < 0.002, Fisher Exact
Statistical Analysis 2: Comparison: q4 Wks vs Placebo; Test type: Superiority or Other; p = 0.200, Fisher Exact

3. Secondary Outcome: Percentage of Subjects With Gout Flare Per 3-month Period
Description: Percent of participants reporting a gout flare during Months 1-3 and Months 4-6. Denominator during the respective period was based upon number of participants during that period.
Time Frame: Months 1-3 and Months 4-6
Population: Number analyzed in each period was based upon number of participants remaining in study during the assessed treatment period: 85/84/43 in Months 1-3 and 69/69/43 in Months 4-6
Measure: Number; unit: Percent subjects reporting flares
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 85 | 84 | 43
Percent subjects reporting flares
  Months 1-3 | 75 | 81 | 54
  Months 4-6 | 41 | 56 | 67
Statistical Analysis 1: Comparison: q2 Wks vs Placebo; % of pegloticase q2 participants reporting flares compared to placebo pts during Months 4-6 treatment period; Test type: Superiority or Other; p = 0.007, Fisher Exact
Statistical Analysis 2: Comparison: q4 Wks vs Placebo; % of pegloticase q4 participants reporting flares compared to placebo pts during Months 4-6 treatment period; Test type: Superiority or Other; p = 0.321, Fisher Exact

4. Secondary Outcome: Change in Number of Swollen Joints
Description: Change from Baseline to Month 6 (or last observation carried forward)in number of swollen joints per subject. Values were inputed using last observation carried forward analysis for subjects who did not complete the studies.
Time Frame: Baseline and Final Visit (Month 6 or LOCF)
Population: All ITT participants with baseline and at least one post-baseline assessment were included in analysis. LOCF was used for participants dropping out early.
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 78 | 77 | 43
Swollen joints | -5.5 (10.47) | -5.1 (7.83) | -2.6 (11.64)
Statistical Analysis 1: Comparison: q2 Wks vs Placebo; Test type: Superiority or Other; p = 0.166, t-test, 2 sided
Statistical Analysis 2: Comparison: q4 Wks vs Placebo; Test type: Superiority or Other; p = 0.170, t-test, 2 sided

5. Secondary Outcome: Change in Number of Tender Joints
Description: Change from Baseline to Month 6 (or last observation carried forward) in number of tender joints per participant
Time Frame: Baseline and Final Visit (Month 6 or LOCF)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 78 | 77 | 43
Tender joints | -7.4 (11.95) | -6.1 (10.64) | -1.2 (12.30)
Statistical Analysis 1: Comparison: q2 Wks vs Placebo; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 2: Comparison: q4 Wks vs Placebo; Test type: Superiority or Other; p = 0.024, t-test, 2 sided

6. Secondary Outcome: Change in Patient Reported Outcomes of Pain, Physical Function and Quality of Life
Description: Health Assessment Questionnaire(HAQ: VAS pain scale where 0 (no pain)-100 (severe pain); HAQ disability index (HAQ-DI) on a scale from 0(no disability) to 3 (completely disabled), and a unit change of > or =0.22 is considerd a mimimal clinically important difference(MCID). SF-36 Physical Component Summary Score (SF36-PCS), a composite score where 0 is the worst score and 100 the best possible, and where a change of > or =2.5 units in the PCS is considered a MCID.
Time Frame: Baseline to Final Visit (Month 6 or LOCF)
Population: Number of participants analyzed was based upon the number who had baseline and at least one follow-up assessment, with the final visit for each subject included (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | q2 Wks | q4 Wks | Placebo
Number analyzed (Participants) | 77 | 77 | 43
Units on a scale
  HAQ-VAS Pain | -11.4 (33.8) | -6.9 (27.0) | 1.4 (30.0)
  HAQ-DI | -0.22 (0.64) | -0.20 (0.55) | 0.0 (0.41)
  SF-36 PCS | 4.4 (9.4) | 4.9 (8.5) | -0.3 (9.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | q2 Wks | q4 Wks | Placebo
Serious Adverse Events (participants affected / at risk) | 20/85 | 19/84 | 5/43
Other Adverse Events (participants affected / at risk) | 69/85 | 79/84 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | q2 Wks (N=85) | q4 Wks (N=84) | Placebo (N=43)
Infusion Related Reaction (General disorders) | 4 (4) | 7 (7) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedoma Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised Infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Necrotising Fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perianal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphyloccal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myopathy Steroid (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gatrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Chronic Lymphocytic Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea Exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | q2 Wks (N=85) | q4 Wks (N=84) | Placebo (N=43)
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 4 | 9
Urinary Tract Infection (Infections and infestations) | 6 | 5 | 3
Nasopharyngitis (Infections and infestations) | 6 | 4 | 1
Localised Infection (Infections and infestations) | 2 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 15 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 14 | 8
Nausea (Gastrointestinal disorders) | 10 | 6 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5 | 1
Constipation (Gastrointestinal disorders) | 5 | 2 | 2
Oedema Peripheral (General disorders) | 9 | 11 | 6
Fatigue (General disorders) | 5 | 6 | 4
Chest Pain (General disorders) | 4 | 4 | 1
Pain (General disorders) | 4 | 4 | 2
Pyrexia (General disorders) | 1 | 5 | 1
Asthenia (General disorders) | 2 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Headache (Nervous system disorders) | 8 | 9 | 4
Dizziness (Nervous system disorders) | 3 | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 0 | 1
Blood Glucose Increased (Investigations) | 4 | 2 | 1
Blood Pressure Increased (Investigations) | 0 | 6 | 0
Insomnia (Psychiatric disorders) | 5 | 8 | 4
Depression (Psychiatric disorders) | 3 | 4 | 4
Hypertension (Vascular disorders) | 2 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 4
Tachycardia (Cardiac disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multicenter publication is to be generated before any individual PI publishes on the results. If multicenter publication is not completed within 18 months from the date of completion, then PI can publish individual results from the Study. Sponsor can review results prior to public release and embargo for no more than 90 days. Sponsor can request removal of Confidential Information only.